CLINICAL TRIAL: NCT05564156
Title: Development and Evaluation of Clinical Pharmacy Services in Respiratory Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Muhammed Yunus BEKTAY, Principal Investigator, Asistant Professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pharm. Role Resp. Disease Ward
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Pneumonia; COPD Asthma; COPD Exacerbation
Keywords: Clinical Pharmacist; Drug-Related Problems; Chest-Diseases; Cognitive Pharmacy Services
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): In the control group; No intervention will be made by the investigators in this group. The participant will take standard treatment. Participant's length of stay in hospital, suitability of antibiotics used, development of microbial resistance, Antibiotic related nephrotoxicity due to infection, mortality data due to infection will be recorded, hospitalization will be questioned within 30 days after the patient is discharged, and a drug consensus report will be created, drug-related problems will be determined, and a pharmacoeconomic evaluation of all possible outcomes will be made. Evaluations will be recorded, but the investigators will take no action.
- Intervention Group (Experimental): In the intervention group; The participant will take standard treatment and the clinical pharmacist services such as drug reconciliation by the investigators, medication review (Identification of drug-related problems, detection of possible unsuitable drugs), quality of life measurement, antibiotic selection, drug suitability, dose and route of administration advice, and concomitant medications are included. Suggestions will be made by the investigators to physicians about the solution to drug-related problems.
  Participants' length of hospital stay, suitability of antibiotics, development of microbial resistance, antibiotic-related nephrotoxicity due to infection, and mortality numbers due to infection will be recorded, hospitalization will be questioned within 30 days after discharge. The investigators will create a drug consensus report, drug-related problems will be determined, and a pharmacoeconomic evaluation of all possible outcomes will be accomplished by investigators.
  Interventions: Behavioral: Intervention groups

INTERVENTIONS:
Behavioral: Intervention groups — The drugs used by the participants within 24-48 hours after hospitalization were recorded. In the case of new prescribing, the recommendations made by the investigators to the physician are recorded in intervention group. The medication reconciliation report will be evaluated before the discharge of the participants and possible omissions discussed with the physician in charge. A detailed medication review will be accomplished by the investigators during the hospitalization of the participants.
  Arms: Intervention Group

SUMMARY:
Clinical pharmacists in the healthcare system are experts in therapeutics and the use of drugs. They routinely provide medication reviews and recommendations to patients and healthcare professionals. Clinical pharmacists are a scientifically valid source of information and give advice on the safe and appropriate use of medicines and pharmacoeconomics. Clinical pharmacist researchers produce, distribute and apply new information that contributes to improving health and quality of life. Thus, it is ensured that many of the drug treatment errors that occur after inappropriate therapeutic decisions are made at the point of prescribing are prevented

In this investigation, the effects of clinical pharmacists on respiratory would be investigated. This research area will cover lower respiratory tract infections and chronic lung disease exacerbations with ICD-10 codes J05, J9-22, J40-47, J69, J85 -J86. In this study, two groups, control and intervention groups, were identified. In the control group; There will be no intervention done by the Clinical Pharmacist. Hospital stay, antimicrobial suitability, microbial resistance development, antimicrobial induced nephrotoxicity, infection-related mortality, pharmacoeconomic evaluation, re-hospitalization within 30 days after discharged, medication reconciliation report will be created, patients will be monitored for the detection and management of drug-related problems will be recorded in both control and intervention groups. In the intervention group; recommendations will be given to the physicians by the Clinical Pharmacist on the selection of antibiotics, drug suitability, dosage and route of administration advice, and determination of drug-related problems related to drugs used simultaneously.

DETAILED DESCRIPTION:
The literature shows the benefit of including the pharmacist in microbiological test review and follow-up. The inclusion of a pharmacist in antibiotic management processes can result in the more reasonable use of antimicrobial agents and more efficient monitoring with patients and/or caregivers. Healthcare policymakers and administrators who evaluate processes to increase efficiency and improve care for patients suspected of discharged infections should examine the effectiveness of clinical pharmacists in the CAP.

Urgent action is needed to tackle the growing resistance threat. Antimicrobial stewardship programs (AYP) have resulted in slowing down antimicrobial resistance and improving antimicrobial prescribing practices that can maintain existing antimicrobial treatments. The CDC and Joint Commission have published recommendations and standards for the conduct of antimicrobial management in both inpatient and outpatient treatment. Although the main principles of the program of antimicrobial management have been established for over a decade, AYPs are constantly evolving, and improving program efficiency brings new approaches to patient care. Although it is one of the main goals of antimicrobial management, the direct effects of AYP interventions on reducing antimicrobial resistance are often immeasurable and multi-factorial. Therefore, interventions aimed at minimizing the use of inappropriate antibiotics, including unnecessary and insufficient use, are often used to measure the effect of AYPs on resistance.

Clinical pharmacists in the healthcare system are experts in therapeutics and the use of drugs. They routinely provide medication reviews and recommendations to patients and healthcare professionals. Clinical pharmacists are a scientifically valid source of information and give advice on the safe and appropriate use of medicines and pharmacoeconomics. Clinical pharmacist researchers produce, distribute and apply new information that contributes to improving health and quality of life.

Clinical pharmacists care about patients in all healthcare areas. They do not only provide clinical services, but they also provide care to their patients and they can perform this application in any application environment. In other words, clinical pharmacists interact and observe directly with the patient. Also, managing treatment directly in patient care settings is particularly important as it reinforces the existing definitions of the term "clinical". In addition, this specialization is used proactively to provide and advance rational drug therapy. Thus, it is ensured that many of the drug treatment errors that occur after inappropriate therapeutic decisions are made at the point of prescribing are prevented.

In this study, two groups, control and intervention groups, were identified. In the control group; There will be no intervention done by the Clinical Pharmacist. Hospital stay, antimicrobial suitability, microbial resistance development, antimicrobial induced nephrotoxicity, infection-related mortality, pharmacoeconomic evaluation, re-hospitalization within 30 days after discharged, medication reconciliation report will be created, patients will be monitored for the detection and management of drug-related problems will be recorded in both control and intervention groups. In the intervention group; recommendations will be given to the physicians by the Clinical Pharmacist on the selection of antibiotics, drug suitability, dosage and route of administration advice, and determination of drug-related problems related to drugs used simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Having any of the J05, J9-22, J40-47, J69, J85-J86 diagnoses specified in the ICD-10 guideline,
* Patients hospitalized due to respiratory tract infection and using antibiotic drugs,
* Being 18 years or older,
* Having signed the written consent form to participate in the study.

Exclusion Criteria:

* The consent form is not approved,
* Not having the necessary cognitive abilities,
* Being under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of suggested intervention | Immediately after the intervention
  Acceptance rate of suggested intervention
Length of hospital stay | Immediately after the discharge of the participant
  Length of hospital stay
30-day readmission | 30 day after the intervention/after the discharge of the each participant
  Readmission within 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Sancar, Prof. Dr., Principal Investigator — Marmara University, Department of Clinical pharmacy
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)